CLINICAL TRIAL: NCT04060706
Title: Hamlet-RT: Heuristics, Algorithms and Machine Learning: Evaluation & Testing in Radiation Therapy
Brief Title: Heuristics, Algorithms and Machine Learning: Evaluation & Testing in Radiation Therapy
Acronym: Hamlet rt
Status: Recruiting | Type: Observational
Sponsor: CCTU- Cancer Theme (Other)
Collaborators: University of Cambridge (Other); Microsoft Research (Industry)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, Dr. Raj Jena, Chief Investigator, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: Hamlet.rt
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Cancer
Keywords: Radiotherapy; Image-guided; Head & Neck; Brain; Lung; Prostate; Adults
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Prostate Cancer: Adults suitable for radical image-guided radiotherapy for their Prostate cancer, approximately 170 patients Components from RTOG, LENT SOM(A), RMH symptom scale and UCLA PCI (prostate cancer index) questionnaires will be used.
  Interventions: Radiation: Radical Image-Guided Radiotherapy
- Head & Neck Cancer: Adults suitable for radical image-guided radiotherapy for their Head & Neck cancer, approximately 140 patients. Components from CTCAE v3, LENT SOM(A), EORTC QLQ H+N35 & Modified xerostomia questionnaires will be used.
  Interventions: Radiation: Radical Image-Guided Radiotherapy
- Central Nervous System Tumours: Adults suitable for radical image-guided radiotherapy for their CNS tumour, as many patients recruited as possible. Components from RTOG, LENT SOM(A), Folstein mini mental state examination & Generalised activites of daily living scale (G-ADL) questionnaires will be used.
  Interventions: Radiation: Radical Image-Guided Radiotherapy
- Lung Cancer: Adults suitable for radical image-guided radiotherapy for their Lung cancer, as many patients recruited as possible. Components from RTOG & LENT SOM(A) questionnaires will be used.
  Interventions: Radiation: Radical Image-Guided Radiotherapy

INTERVENTIONS:
Radiation: Radical Image-Guided Radiotherapy — Questionnaires administered will monitor the clinical toxicity experienced by each patient up to 5 years post radiotherapy

SUMMARY:
The Hamlet.rt study is a prospective data collection and patient questionnaire study for patients undergoing image-guided radiotherapy with curative intent.

The aim of the study is to use novel machine learning and mathematical techniques to build a model that can predict the risk of significant side effects from radiotherapy treatment for an individual patient: using calculations of normal tissue dose from radiotherapy treatment planning and patient baseline characteristics derived from image and non-image data, continuously updated as the patient is reviewed both during and after treatment.

A secondary goal of the project is to facilitate research in machine learning and medical image processing for radiation therapy through the creation of a discoverable and shared data resource for research use.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or Female
* Aged 18 years or older
* Diagnosed with primary prostate cancer, head and neck cancer, lung cancer, or brain tumour
* Treated with curative intent
* Suitable for radical image guided radiotherapy
* WHO ECOG performance status 0 or 1
* Expected survival of 18 months or more

Exclusion Criteria:

* Participant is not willing or able to complete the protocol-stated requirements of the study, e.g. accessing & completing web-based long-term follow-up questionnaires.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults suitable for radical image-guided radiotherapy with Prostate, Head & Neck, Brain, or Lung Cancer. The variation in conditions is based on the requirements of Machine Learning algorithms requiring high levels of clinical applicability, which depends on the quality and quantity of the input data available. The input data set therefore should adequately encompass the variation in anatomy encountered in the population.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2019-09-11 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Machine Learning Modelling | 8 years from FPFV
  Characterise machine learning models for the four disease sites. Developing machine learning algorithms for autosegmentation of normal tissue anatomy, and to extend machine learning algorithms to identify and segment normal tissue structures in cone beam CT images, and to utilise the ML segmentations to evaluate image signatures correlated with treatment toxicity
Predictive Modelling | 8 years from FPFV
  Predict performance matches with published techniques. Combining the machine learning models in outcome 1, with pre-treatment assessment data and on-treatment quantitative assessments in outcome 3 for the construction and evaluation of a predictive mathematical model
Clinical Toxicity Evaluation | 8 years from FPFV
  Evaluation of the clinical toxicity experienced by each patient up to 5 years post radiotherapy to inform the predictive models in outcome 2

CONTACTS AND LOCATIONS:
Overall Officials: Raj Dr. Jena, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust & the University of Cambridge; Suzanne Miller, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust; Amy Bates, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided